CLINICAL TRIAL: NCT05819320
Title: Pattern of Mucocutaneous Manifestations in Patients With Chronic Kidney Disease in New Vally and Assuit (Hospital Based Study) .
Brief Title: Mucocutaneous Manifestations in Patients With Chronic Kidney Disease inNewVally and Assuit;Hospital Based Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Hassan Mohammed Ahmed, Dr Marwa Hassan Mohammed, Assiut University
Other Study IDs: skin manifestations in CKD
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases; Manifestation, Skin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Skin Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ALdakhla general hospital patients: patterns of mucocutaneous manifestations and their correlation with the different stages of Chronic Kidney Disease in renal unit of internal medicine of Eldakhla general hospital in New Vally
  Interventions: Other: observe pattern of mucocutaneous manifestations in chronic kidney disease patients
- Assuit University hospital adult renal unit: patterns of mucocutaneous manifestations and their correlation with the different stages of Chronic Kidney Disease in renal unit of internal medicine of Assuit University hospital (adult renal unit ) .
  Interventions: Other: observe pattern of mucocutaneous manifestations in chronic kidney disease patients
- Assuit University hospital pediatric renal unit: patterns of mucocutaneous manifestations and their correlation with the different stages of Chronic Kidney Disease in renal unit of internal medicine of Assuit University hospital (pediatric renal unit ).
  Interventions: Other: observe pattern of mucocutaneous manifestations in chronic kidney disease patients

INTERVENTIONS:
Other: observe pattern of mucocutaneous manifestations in chronic kidney disease patients — 1. To study the patterns of mucocutaneous disorders in Chronic Kidney Disease patients .
  2. Comparison of the patterns of mucocutaneous manifestations and their correlation with the different stages of Chronic Kidney Disease

SUMMARY:
1. To study the patterns of mucocutaneous disorders in Chronic Kidney Disease patients in Eldakhla General Hospital, New Valley and in Assiut University hospital .
2. Comparison of the patterns of mucocutaneous manifestations and their correlation with the different stages of Chronic Kidney Disease in renal unit of internal medicine of Eldakhla general hospital in New Vally and pediatric and adult renal units of Assuit university hospital .

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is defined as abnormalities of kidney structure or function , present for > 3 months , with implications for health . chronic kidney disease is classified based on cause , Glomerular Filtration Rate category (G1-G5) , and Albuminuria category ( A1-A3) , abbreviated as CGA . (Michel et al.,2023).

Chronic kidney disease (CKD) affects up to 13% of the population and may progress to kidney failure and death. Some risk factors for chronic kidney disease are well known such as high blood pressure and diabetes. There is some evidence that inflammatory skin diseases such as eczema and psoriasis may also increase the risk of chronic kidney disease . (Schonmann et al.,2021).

Skin serves as the mirror of underlying systemic problems. The early diagnosis of subtle cutaneous clinical pointers often helps in identifying renal disorders, obviating the delay in diagnosis and treatment. Cutaneous changes can be observed from the beginning of renal impairment until the evolution to terminal stage . ( Vivek et al,2021) Most patients with severe chronic kidney disease progress to end stage renal disease (ESRD). Cutaneous manifestations are common in all stages of chronic kidney disease particularly towards end stage renal disease . (Rattan et al.,2018).

The prevalence of chronic kidney disease is increasing, and the incidence and prevalence of associated skin diseases will also increase. Their early recognition and treatment to reduce morbidity and mortality are essential . (Timur et al,2014) Many factors are involved in the pathogenesis of the cutaneous manifestations of end stage renal disease , including electrolyte imbalance, buildup of uremic substances, and comorbid disease (Goldman et al,2012).

There are two main categories of the cutaneous manifestations of chronic kidney diseases: nonspecific and specific.

Nonspecific manifestations include pruritus, skin color changes, xerosis, and half-and-half nails. Specific manifestations include acquired perforating dermatosis, bullous dermatoses, metastatic calcification, and nephrogenic systemic fibrosis. (Goldman et al,2012).

The pattern of mucocutaneous manifestations of chronic kidney disease in Eldakhla, the New Valley, Egypt, are not studied before.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic kidney disease attending the renal unit of internal medicine of Eldakhla General hospital, New Vally ,and Assiut University hospital will be included in this study within two years and will be examined for any skin manifestations and mucocutaneous findings.

Exclusion Criteria:

- Human immunodeficiency (HIV) affected persons, renal transplant recipients, and patients with acute renal failure, hepatobiliary, pancreatic, or thyroid disorders, cutaneous or systemic malignancies will be excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with chronic kidney disease attending the renal unit of internal medicine of Eldakhla General hospital, New Vally ,and Assiut University hospital will be included in this study .
  Detailed medical history, clinical examination and investigations which support the diagnosis will be recorded including: urine analysis, CBC, Blood urea, creatinine , x- ray, arterial blood gases , abdominal sonography ,serum electrolytes, multislice CT KUB , Demsa scan ......etc .
  Potassium hydroxide (KOH) mounts, skin biopsy, Gram's, and Giemsa staining, and bacterial or fungal cultures will be performed when we need.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
study the patterns of mucocutaneous disorders in Chronic Kidney Disease patients in Eldakhla General Hospital, New Valley and in Assiut University hospital | Base line
  Comparison of the patterns of mucocutaneous manifestations and their correlation with the different stages of Chronic Kidney Disease in renal unit of internal medicine of Eldakhla general hospital in New Vally and pediatric and adult renal units of Assuit university hospital .

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Samir sayed, Study Director — Supervisor; Eman Mohammed kamal Elsayed Yousef, Study Director — Supervisor; Marwa Hassan Mohammed, Principal Investigator — Investigator

REFERENCES:
- [Background] Schonmann Y, Mansfield KE, Mulick A, Roberts A, Smeeth L, Langan SM, Nitsch D. Inflammatory skin diseases and the risk of chronic kidney disease: population-based case-control and cohort analyses. Br J Dermatol. 2021 Oct;185(4):772-780. doi: 10.1111/bjd.20067. Epub 2021 Jun 6. PMID 33730366
- [Background] Rashpa RS, Mahajan VK, Kumar P, Mehta KS, Chauhan PS, Rawat R, Sharma V. Mucocutaneous Manifestations in Patients with Chronic Kidney Disease: A Cross-sectional Study. Indian Dermatol Online J. 2018 Jan-Feb;9(1):20-26. doi: 10.4103/idoj.IDOJ_160_17. PMID 29441293
- [Background] Galperin TA, Cronin AJ, Leslie KS. Cutaneous manifestations of ESRD. Clin J Am Soc Nephrol. 2014 Jan;9(1):201-18. doi: 10.2215/CJN.05900513. Epub 2013 Oct 10. PMID 24115194
- [Background] Goel V, Sil A, Das A. Cutaneous Manifestations of Chronic Kidney Disease, Dialysis and Post-Renal Transplant: A Review. Indian J Dermatol. 2021 Jan-Feb;66(1):3-11. doi: 10.4103/ijd.IJD_502_20. PMID 33911288